CLINICAL TRIAL: NCT01187355
Title: SiH MPDS FID 114675A Compared to Renu Fresh MPS in Symptomatic Contact Lens Wearers
Brief Title: Alcon Multi-Purpose Disinfecting Solution Versus Renu Fresh Multi-Purpose Solution in Symptomatic Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: C-09-074
Record Dates: First submitted 2010-08-20; First posted 2010-08-24 (Estimated); Results first posted 2012-07-30 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-06

CONDITIONS: Symptomatic Contact Lens Wearers
Keywords: Symptomatic, Contact lens care; Multi-purpose solution
MeSH Terms: interventions — Contact Lenses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alcon MPDS (Experimental): MPDS used for 30 days as specified in protocol for contact lens care.
  Interventions: Device: FID 114675A Multi-Purpose Disinfecting Solution (MPDS); Device: Contact lenses
- renu fresh MPS (Active Comparator): MPS used for 30 days as indicated for contact lens care.
  Interventions: Device: renu fresh Multi-Purpose Solution (MPS); Device: Contact lenses

INTERVENTIONS:
Device: FID 114675A Multi-Purpose Disinfecting Solution (MPDS) — Investigational multi-purpose disinfecting solution used by subjects as specified in use instructions provided for the care of study contact lenses, 30 days.
  Arms: Alcon MPDS
Device: renu fresh Multi-Purpose Solution (MPS) — Commercially available multi-purpose solution used by subjects as indicated for care of study contact lenses, 30 days.
  Other Names: renu® fresh™ Multi-Purpose Solution
  Arms: renu fresh MPS
Device: Contact lenses — Contact lenses per subject's habitual brand and power worn for 30 days on a daily wear basis.

SUMMARY:
The purpose of this study is to compare two contact lens care solutions in symptomatic wearers of silicone hydrogel contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic silicone hydrogel contact lens wearers who wear their lenses daily wear (i.e., disinfect lenses every night).
* Vision correctable to 20/30 or better with contact lenses.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Sensitivity to multi-purpose solutions.
* Use of any topical ocular OTC or prescribed topical ocular medications.
* History (6 months) or current ocular infections or ocular inflammatory events.
* Ocular surgery within the past year.
* Medical condition or use of medications that cause ocular side effects.
* Participation in any investigational study within the past 30 days.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 591 (Actual)
Dates: Start 2010-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited and enrolled from 42 US study centers.
Pre-assignment Details: The Participant Flow Chart includes all randomized patients: 591. Baseline characteristics are presented for all subjects who received test article and had at least one on-regimen study visit: 578.
Groups:
- Alcon MPDS: Multi-purpose disinfecting contact lens solution
- Renu Fresh MPS: Multi-purpose contact lens solution
Period: Overall Study
Arm/Group | Alcon MPDS | Renu Fresh MPS
Started | 294 | 297
Completed | 276 | 277
Not Completed | 18 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alcon MPDS | Renu Fresh MPS | Total
Number analyzed (Participants) | 288 | 290 | 578
Age Continuous [Mean (Standard Deviation); unit: years] | 34.5 (11.43) | 34.0 (11.24) | 34.3 (11.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 209 | 212 | 421
  Male | 79 | 78 | 157

OUTCOME MEASURES:

1. Primary Outcome: Likert Statement: When I Use This Solution, I Can Comfortably Wear my Lenses.
Description: As interpreted and reported by the subject on a questionnaire as a single, retrospective evaluation of the last three days of wearing experience. A 5-point Likert scale was used, where 1=strongly disagree, 2=disagree; 3=neither disagree nor agree; 4=agree; 5=strongly agree.
Time Frame: Day 30
Population: All enrolled and dispensed subjects with an on-regimen follow-up visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Alcon MPDS | Renu Fresh MPS
Number analyzed (Participants) | 276 | 277
Units on a scale | 3.9 (0.92) | 3.8 (1.05)

2. Secondary Outcome: Likert Statement: When I Use This Solution, My Lenses Are Comfortable From Morning Until Evening.
Description: as for outcome 1
Time Frame: Day 30
Population: All enrolled and dispensed subjects with an on-regimen follow-up visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Alcon MPDS | Renu Fresh MPS
Number analyzed (Participants) | 276 | 276
Units on a scale | 3.3 (1.12) | 3.2 (1.21)

3. Secondary Outcome: Likert Statement: When I Use This Solution, I Forget I am Wearing my Lenses.
Description: as for outcome 1
Time Frame: Day 30
Population: All enrolled and dispensed subjects with an on-regimen follow-up visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Alcon MPDS | Renu Fresh MPS
Number analyzed (Participants) | 276 | 277
Units on a scale | 3.2 (1.13) | 3.1 (1.15)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study: 5 months, 2 weeks, 1 day.
Description: This reporting group includes all subjects enrolled and dispensed test article.
Arm/Group | Alcon MPDS | Renu Fresh MPS
Serious Adverse Events (participants affected / at risk) | 1/292 | 1/297
Other Adverse Events (participants affected / at risk) | 0/292 | 0/297
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alcon MPDS (N=292) | Renu Fresh MPS (N=297)
Schizoaffective Disorder Bipolar Type (Psychiatric disorders) | 1 (1) | 0 (0)
Abortion Spontaneous (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.